CLINICAL TRIAL: NCT01760447
Title: A Pooled Analysis of the Safety and Efficacy of MK-0431A and MK-0431A XR in Pediatric Patients With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Metformin Therapy (Alone or in Combination With Insulin)
Brief Title: A Pooled Analysis of the Safety and Efficacy of MK-0431A and MK-0431A XR in Pediatric Participants With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Metformin Therapy (Alone or in Combination With Insulin) (MK-0431A-170/MK-0431A-289)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0431A-289; 2012-004035-23 (EudraCT Number); 2011-002529-23 (EudraCT Number); 2014-003583-20 (EudraCT Number); MK-0431A-170 (Other: Merck Protocol Number); MK-0431A-289 (Other: Merck Protocol Number); CTRI/2012/09/003025 (Registry Identifier: CTRI); NCT01472367 (obsolete NCT alias)
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Results first posted 2020-10-05 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin; Insulin

STUDY DESIGN:
Intervention Model Description: Participants enrolled in protocol MK-0431A-170 were randomized between the arms "Sitagliptin/Metformin" and "Metformin." Participants enrolled in protocol MK-0431A-289 were randomized between the arms "Sitagliptin/Metformin XR" and "Metformin XR."
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants enrolled in protocol MK-0431A-170 were aware that they would receive either sitagliptin and metformin, or metformin. Participants in protocol MK-0431A-289 were aware that they would receive either sitagliptin and metformin XR, or metformin XR.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sitagliptin/Metformin (Experimental): Participants received one tablet of sitagliptin/metformin and one tablet of metformin-placebo, administered twice daily prior to the morning and evening meals, for up to 20 weeks in the base study alone, or for up to 54 weeks if the participant also entered the extension study. Participants in this arm were enrolled in protocol MK-0431A-170.
  Interventions: Drug: Sitagliptin plus metformin; Drug: Placebo to metformin; Drug: Insulin
- Metformin (Placebo Comparator): Participants received one tablet of metformin and one tablet of placebo to sitagliptin/metformin, administered twice daily prior to the morning and evening meals, for up to 20 weeks in the base study alone, or for up to 54 weeks if the participant also entered the extension study. Participants in this arm were enrolled in protocol MK-0431A-170.
  Interventions: Drug: Metformin; Drug: Placebo to sitagliptin plus metformin; Drug: Insulin
- Sitagliptin/Metformin XR (Experimental): Participants received two tablets of sitagliptin/metformin XR and two tablets of metformin XR placebo, administered once daily with a meal, for up to 54 weeks. Participants in this arm were enrolled in protocol MK-0431A-289.
  Interventions: Drug: Sitagliptin plus metformin XR; Drug: Placebo to metformin XR; Drug: Insulin
- Metformin XR (Placebo Comparator): Participants received two tablets of metformin XR and two tablets of placebo to sitagliptin/metformin XR, administered once daily with a meal, for up to 54 weeks. Participants in this arm were enrolled in protocol MK-0431A-289.
  Interventions: Drug: Insulin; Drug: Placebo to sitagliptin plus metformin XR; Drug: Metformin XR

INTERVENTIONS:
Drug: Sitagliptin plus metformin — Participants received 2 tablets daily, one taken with a morning meal and one taken with an evening meal, to provide a total daily dose of 100 mg of sitagliptin and 1000 mg, 1700 mg or 2000 mg of metformin. Dosage of metformin was based on each participant's daily metformin dose prior to enrollment.
  Other Names: MK-0431A
  Arms: Sitagliptin/Metformin
Drug: Placebo to metformin — Participants received 2 tablets daily, one taken with a morning meal and one taken with an evening meal. Each tablet contained placebo to metformin.
  Arms: Sitagliptin/Metformin
Drug: Metformin — Participants received 2 tablets daily, one taken with a morning meal and one taken with an evening meal, to provide a total daily dose of 1000 mg, 1700 mg or 2000 mg of metformin. Dosage was based on each participant's daily metformin dose prior to enrollment.
  Arms: Metformin
Drug: Placebo to sitagliptin plus metformin — Participants received 2 tablets daily, one taken with a morning meal and one taken with an evening meal. Each tablet contained placebo to sitagliptin plus metformin.
  Other Names: Placebo to MK-0431A
  Arms: Metformin
Drug: Sitagliptin plus metformin XR — Participants received 2 tablets daily, both taken together with a meal, to provide a total daily dose of 100 mg of sitagliptin and 1000 mg, 1500 mg or 2000 mg of metformin. Dosage of metformin XR was based on each participant's daily metformin dose prior to enrollment.
  Other Names: MK-0431A XR
  Arms: Sitagliptin/Metformin XR
Drug: Placebo to metformin XR — Participants received 2 tablets daily, both taken together with a meal. Each tablet contained placebo to metformin XR.
  Arms: Sitagliptin/Metformin XR
Drug: Insulin — Participants who met protocol-specific glycemic rescue criteria received insulin as glycemic rescue therapy; participants on background insulin had their insulin dose increased for glycemic rescue. During Weeks 20-54, for participants who were not on background insulin or rescued with insulin during Weeks 0-20 in the "Sitagliptin/Metformin" and "Metformin" arms (protocol MK-0431A-170), and during Weeks 0-54 for participants not on background insulin in the "Sitagliptin/Metformin XR" and "Metformin XR" arms (protocol MK-0431A-289), the type of insulin for glycemic rescue was specified to be insulin glargine.
Drug: Placebo to sitagliptin plus metformin XR — Participants received 2 tablets daily, both taken together with a meal. Each tablet contained placebo to sitagliptin plus metformin XR.
  Other Names: Placebo to MK-0431A XR
  Arms: Metformin XR
Drug: Metformin XR — Participants received 2 tablets daily, both taken together with a meal, to provide a total daily dose of 1000 mg, 1500 mg or 2000 mg of metformin XR. Dosage was based on each participant's daily metformin dose prior to enrollment.
  Arms: Metformin XR

SUMMARY:
The purpose of this study is to assess the effect of the addition of sitagliptin (administered as MK-0431A or MK-0431A XR) relative to the addition of placebo on glycated hemoglobin (A1C), and the safety and tolerability of the addition of sitagliptin, in pediatric participants (ages 10-17 years) with type 2 diabetes mellitus with inadequate glycemic control on metformin therapy (alone or in combination with insulin). The primary hypothesis is that the addition of sitagliptin reduces glycated hemoglobin (A1C) more than the addition of placebo after 20 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* For MK-0431A-170 base study and MK-0431A-289:

  * Has type 2 diabetes mellitus (T2DM)
  * Is on metformin monotherapy (≥1500 mg/day) for ≥12 weeks with glycated hemoglobin (A1C) ≥6.5% and ≤10.0% OR is on stable doses of metformin (≥1500 mg/day) and insulin for ≥12 weeks with an A1C ≥7.0% and ≤10%. NOTE: Participants on a daily dose of metformin greater than or equal to 1000 mg/day, but less than 1500 mg/day may be eligible if there is documentation that higher doses are not tolerated.
  * Participant and a family member or adult closely involved in the daily activities will participate in the participant's treatment and study protocol (i.e., available for telephone calls, study visits and administration of study medication as needed).
  * Male, or female who is unlikely to conceive (non-sterilized, and is not sexually active or agrees to abstain from heterosexual activity or agrees to use an adequate method of contraception) during the study and for 14 days after the last dose of study drug
* For MK-0431A-170 extension protocol:

  * Has completed the P170 base study
  * Participant and a family member or adult closely involved in the daily activities will participate in the participant's treatment and study protocol (i.e., available for telephone calls, study visits and administration of study medication as needed).
  * Male, or female who is unlikely to conceive (non-sterilized, and is not sexually active or agrees to abstain from heterosexual activity or agrees to use an adequate method of contraception) during the study and for 14 days after the last dose of study drug

Exclusion Criteria:

* For MK-0431A-170 base study and MK-0431A-289:

  * Has type 1 diabetes mellitus
  * Has monogenic diabetes or secondary diabetes
  * Has symptomatic hyperglycemia and/or moderate to large ketonuria and/or positive test for ketonemia, requiring immediate initiation of another antihyperglycemic agent
  * Has previously taken a dipeptidyl peptidase IV (DPP-4) inhibitor (such as sitagliptin, vildagliptin, alogliptin, saxagliptin, or linagliptin) or glucagon-like peptide-1 (GLP-1) receptor agonist (such as exenatide or liraglutide)
  * Is on or likely to require treatment for ≥2 consecutive weeks or repeated courses of corticosteroids (inhaled, nasal and topical corticosteroids are permitted)
  * Has undergone a surgical procedure within 4 weeks of study participation or has planned major surgery during the study
  * History of congenital heart disease or cardiovascular disease other than hypertension
  * History of active liver disease (other than non-alcoholic steatosis), including chronic active hepatitis B or C, primary biliary cirrhosis, or symptomatic gallbladder disease
  * Active neuropathy (such as nephrotic syndrome or glomerulonephritis)
  * Chronic myopathy, mitochondrial disorder or a progressive neurological or neuromuscular disorder
  * Human immunodeficiency virus (HIV)
  * Hematological disorder (such as aplastic anemia, thrombocytopenia, myeloproliferative or myelodysplastic syndromes)
  * Is currently being treated for hyperthyroidism or is on thyroid hormone therapy and has not been on a stable dose for at least 6 weeks
  * History of malignancy for ≤5 years prior to study participation, except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer
  * History of idiopathic acute pancreatitis or chronic pancreatitis
  * History of recreational or illicit drug use, or of alcohol abuse or dependence (within the past year)
  * Has donated blood products or has had phlebotomy of >10% of estimated total blood volume within 8 weeks of study participation, or intends to donate blood products or receive blood products within the projected duration of the study
  * Is pregnant or breast-feeding, or is expecting to conceive or donate eggs during the study, including 14 days following the last dose of study drug
* For MK-0431A-170 extension protocol:

  * Participant meets a study medication discontinuation criterion at the last visit of the MK-0431A-170 base study (Week 20)
  * Has taken the last dose of study medication for the MK-0431A-170 base study more than 14 days prior to Extension Visit 1
  * Has initiated another oral antihyperglycemic agent
  * Participant does not agree to refrain from participating in any other double-blind interventional study while participating in the P170 extension study

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 223 (Actual)
Dates: Start 2011-12-07 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Jalaludin MY, Deeb A, Zeitler P, Garcia R, Newfield RS, Samoilova Y, Rosario CA, Shehadeh N, Saha CK, Zhang Y, Zilli M, Scherer LW, Lam RLH, Golm GT, Engel SS, Kaufman KD, Shankar RR. Efficacy and safety of the addition of sitagliptin to treatment of youth with type 2 diabetes and inadequate glycemic control on metformin without or with insulin. Pediatr Diabetes. 2022 Mar;23(2):183-193. doi: 10.1111/pedi.13282. Epub 2021 Dec 20. PMID 34779103

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited participants in clinics/clinical offices in 28 countries.
  One participant who was randomized to the arm "Sitagliptin/Metformin" withdrew prior to treatment, then was re-randomized into the study. Only the second randomization is counted for Participant Flow and All-Cause Mortality, so this participant is not counted twice.
Pre-assignment Details: The Pre-Assignment Period included a one-week single-blind placebo run-in prior to randomization during which participants received metformin with sitagliptin/metformin placebo or metformin XR with sitagliptin/metformin XR placebo each day.
Period: Weeks 0-20
Arm/Group | Sitagliptin/Metformin | Metformin | Sitagliptin/Metformin XR | Metformin XR
Started | 62 (The first randomization for the participant who withdrew and re-randomized is not counted in the 62.) | 62 | 47 | 51
Treated | 62 | 62 | 45 | 51
Completed | 59 | 62 | 42 | 47
Not Completed | 3 | 0 | 5 | 4
Not completed — Consent withdrawn by Parent/Guardian | 0 | 0 | 1 | 3
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 1
Not completed — Randomized but not treated | 0 | 0 | 2 | 0
Period: Weeks 20-54
Arm/Group | Sitagliptin/Metformin | Metformin | Sitagliptin/Metformin XR | Metformin XR
Started | 28 (MK-0431A-170 added Weeks 20-54 via amendment, but not all participants were eligible for this period) | 30 (MK-0431A-170 added Weeks 20-54 via amendment, but not all participants were eligible for this period) | 42 | 47
Completed | 25 | 28 | 39 | 43
Not Completed | 3 | 2 | 3 | 4
Not completed — Consent withdrawn by Parent/Guardian | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: The baseline characteristics data are presented for all treated participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin/Metformin | Metformin | Sitagliptin/Metformin XR | Metformin XR | Total
Number analyzed (Participants) | 62 | 62 | 45 | 51 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.4 (2.2) | 13.9 (1.8) | 14.8 (1.9) | 14.9 (1.6) | 14.4 (1.9)
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0 | 0 | 0
  Children (2-11 years) | 10 | 7 | 3 | 1 | 21
  Adolescents (12-17 years) | 52 | 55 | 42 | 50 | 199
  Adults (18-64 years) | 0 | 0 | 0 | 0 | 0
  From 65-84 years | 0 | 0 | 0 | 0 | 0
  85 years and over | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 40 | 32 | 32 | 145
  Male | 21 | 22 | 13 | 19 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 23 | 11 | 20 | 77
  Not Hispanic or Latino | 35 | 36 | 29 | 28 | 128
  Unknown or Not Reported | 4 | 3 | 5 | 3 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 3 | 9 | 13
  Asian | 21 | 22 | 15 | 6 | 64
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 0 | 2
  Black or African American | 2 | 2 | 2 | 4 | 10
  White | 24 | 23 | 22 | 27 | 96
  More than one race | 14 | 13 | 3 | 5 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Glycated Hemoglobin (A1C) [Mean (Standard Deviation); unit: Percentage] — Glycated hemoglobin (A1C) is a blood marker used to report average blood glucose levels over prolonged periods of time. Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100.
  Percentage | 8.02 (1.22) | 8.13 (1.08) | 7.87 (0.94) | 7.97 (1.05) | 8.0 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in A1C at Week 20
Description: Glycated hemoglobin (A1C) is a blood marker used to report average blood glucose levels over prolonged periods of time. Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100. Mean change from baseline at Week 20 was estimated from a longitudinal data analysis model.
Time Frame: Baseline and Week 20
Population: The analysis population includes all randomized participants who received ≥1 dose of study medication and who had at least 1 measurement of A1C. As defined in the protocols, these analyses were conducted in participants pooled from protocols MK-0431A-170 and MK-0431A-289, pooled according to receipt of experimental drug or placebo comparator.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of glycated hemoglobin
Groups:
- Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled: This reporting group contains the pooled population of treated participants from the experimental-drug groups "Sitagliptin/Metformin" (from protocol MK-0431A-170) and "Sitagliptin/Metformin XR" (from protocol MK-0431A-289).
- Metformin and Metformin XR Pooled: This reporting group contains the pooled population of treated participants from the placebo groups "Metformin" (from protocol MK-0431A-170) and "Metformin XR" (from protocol MK-0431A-289).
Arm/Group | Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled | Metformin and Metformin XR Pooled
Number analyzed (Participants) | 107 | 113
Percentage of glycated hemoglobin | -0.58 [-0.94 to -0.22] | -0.09 [-0.43 to 0.26]
Statistical Analysis 1: Comparison: Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled vs Metformin and Metformin XR Pooled; The Least Squares (LS) Mean for the arm "Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled" is compared against that of "Metformin and Metformin XR Pooled."; Test type: Superiority; p = 0.018, Mixed Models Analysis; Least Squares Mean Difference = -0.49, 95% CI 2-sided [-0.90 to -0.09]

2. Primary Outcome: Number of Participants Who Experienced ≥1 Adverse Event During Weeks 0-20
Description: The number of participants experiencing ≥1 adverse event during Weeks 0-20 was reported. An adverse event is defined as any untoward medical occurrence in a person administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to Week 20
Population: The analysis population includes all randomized participants who received ≥1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin/Metformin | Metformin | Sitagliptin/Metformin XR | Metformin XR | Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled | Metformin and Metformin XR Pooled
Number analyzed (Participants) | 62 | 62 | 45 | 51 | 107 | 113
Participants | 42 | 46 | 29 | 30 | 71 | 76
Statistical Analysis 1: Comparison: Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled vs Metformin and Metformin XR Pooled; The percentage of participants who experienced ≥1 adverse event for the arm "Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled" is compared against that of "Metformin and Metformin XR Pooled."; Test type: Other; Difference in Percentage = -1.3, 95% CI 2-sided [-13.9 to 11.3] — The Miettinen and Nurminen methodology was used to calculate the difference and 95% confidence interval

3. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to Experiencing an Adverse Event During Weeks 0-20
Description: The number of participants who discontinued from study drug due to an adverse event during Weeks 0-20 was reported. An adverse event is defined as any untoward medical occurrence in a person administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to Week 20
Population: The analysis population includes all randomized participants who received ≥1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin/Metformin | Metformin | Sitagliptin/Metformin XR | Metformin XR | Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled | Metformin and Metformin XR Pooled
Number analyzed (Participants) | 62 | 62 | 45 | 51 | 107 | 113
Participants | 1 | 2 | 2 | 2 | 3 | 4
Statistical Analysis 1: Comparison: Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled vs Metformin and Metformin XR Pooled; The percentage of participants who discontinued study drug due to experiencing an adverse event for the arm "Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled" is compared against that of "Metformin and Metformin XR Pooled."; Test type: Other; Difference in Percentage = -0.5, 95% CI 2-sided [-6.2 to 5.0] — The Miettinen and Nurminen methodology was used to calculate the difference and 95% confidence interval

4. Primary Outcome: Number of Participants Who Experienced ≥1 Adverse Event During Weeks 0-56
Description: The number of participants experiencing ≥1 adverse event during Weeks 0-56 were reported. An adverse event is defined as any untoward medical occurrence in a person administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to approximately Week 56
Population: The analysis population includes all randomized participants who received ≥1 dose of study medication and continued in the study beyond Week 20.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin/Metformin | Metformin | Sitagliptin/Metformin XR | Metformin XR | Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled | Metformin and Metformin XR Pooled
Number analyzed (Participants) | 28 | 30 | 42 | 47 | 70 | 77
Participants | 26 | 27 | 36 | 39 | 62 | 66
Statistical Analysis 1: Comparison: Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled vs Metformin and Metformin XR Pooled; [analysis description as in outcome 2, analysis 1]; Test type: Other; Difference in Percentage = 2.9, 95% CI 2-sided [-8.9 to 14.4] — The Miettinen and Nurminen methodology was used to calculate the difference and 95% confidence interval

5. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to Experiencing an Adverse Event During Weeks 0-54
Description: The number of participants who discontinued from study drug due to an adverse event during Weeks 0-54 was reported. An adverse event is defined as any untoward medical occurrence in a person administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to Week 54
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin/Metformin | Metformin | Sitagliptin/Metformin XR | Metformin XR | Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled | Metformin and Metformin XR Pooled
Number analyzed (Participants) | 28 | 30 | 42 | 47 | 70 | 77
Participants | 1 | 1 | 1 | 3 | 2 | 4
Statistical Analysis 1: Comparison: Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled vs Metformin and Metformin XR Pooled; [analysis description as in outcome 3, analysis 1]; Test type: Other; Difference in Percentage = -2.1, 95% CI 2-sided [-10.1 to 5.8] — The Miettinen and Nurminen methodology was used to calculate the difference and 95% confidence interval

6. Secondary Outcome: Change From Baseline in A1C at Week 54
Description: A1C is a blood marker used to report average blood glucose levels over prolonged periods of time. Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100. Mean change from baseline at Week 54 was estimated from a longitudinal data analysis model.
Time Frame: Baseline and Week 54
Population: The analysis population includes all randomized participants who received ≥1 dose of study medication, had ≥1 measurement of A1C, and continued in the study beyond Week 20. As defined in the protocols, these analyses were conducted in participants pooled from protocols MK-0431A-170 and -289, pooled by receipt of experimental drug or placebo.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of glycated hemoglobin
Arm/Group | Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled | Metformin and Metformin XR Pooled
Number analyzed (Participants) | 70 | 77
Percentage of glycated hemoglobin | 0.35 [-0.48 to 1.19] | 0.73 [-0.08 to 1.54]

7. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 20
Description: Blood glucose was measured on a fasting basis. Mean change from baseline at Week 20 was estimated from a longitudinal data analysis model.
Time Frame: Baseline and Week 20
Population: The analysis population includes all randomized participants who received ≥1 dose of study medication, and who had at least 1 measurement of FPG. As defined in the protocols, these analyses were conducted in participants pooled from protocols MK-0431A-170 and MK-0431A-289, pooled according to receipt of experimental drug or placebo comparator.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled | Metformin and Metformin XR Pooled
Number analyzed (Participants) | 107 | 113
mg/dL | -2.5 [-16.7 to 11.7] | 8.3 [-5.0 to 21.6]
Statistical Analysis 1: Comparison: Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled vs Metformin and Metformin XR Pooled; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.159, Mixed Models Analysis; Least Squares Mean Difference = -10.8, 95% CI 2-sided [-25.9 to 4.3]

8. Secondary Outcome: Change From Baseline in FPG at Week 54
Description: Blood glucose was measured on a fasting basis. Mean change from baseline at Week 54 was estimated from a longitudinal data analysis model.
Time Frame: Baseline and Week 54
Population: The analysis population includes all randomized participants who received ≥1 dose of study medication, had ≥1 measurement of FPG, and continued in the study beyond Week 20. As defined in the protocols, these analyses were conducted in participants pooled from protocols MK-0431A-170 and -289, pooled by receipt of experimental drug or placebo.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled | Metformin and Metformin XR Pooled
Number analyzed (Participants) | 70 | 77
mg/dL | 16.8 [-8.4 to 42.0] | 16.9 [-7.0 to 40.8]

9. Secondary Outcome: Percentage of Participants With A1C at Goal (<7.0%) at Week 20
Description: Glycated hemoglobin (A1C) is a blood marker used to report average blood glucose levels over prolonged periods of time. Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100. Percentage of participants with A1C at goal (<7.0%) at Week 20 was presented.
Time Frame: Week 20
Population: The analysis population includes all randomized participants who received ≥1 dose of study medication. As defined in the protocols, these analyses were conducted in participants pooled from protocols MK-0431A-170 and MK-0431A-289, pooled according to receipt of experimental drug or placebo comparator.
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled | Metformin and Metformin XR Pooled
Number analyzed (Participants) | 107 | 113
Percentage of participants | 43.0 | 31.0
Statistical Analysis 1: Comparison: Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled vs Metformin and Metformin XR Pooled; The percentage of participants with A1C at the A1C goal (<7.0%) in the arm "Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled" is compared against that of "Metformin and Metformin XR Pooled." For estimating the treatment difference, when the A1C result for a participant at Week 20 was not available, a multiple imputation method was used to impute whether the participant had met the goal; Test type: Superiority; p = 0.017, Miettinen and Nurminen; Difference in Percentage = 16.0, 95% CI 2-sided [2.9 to 28.9]

10. Secondary Outcome: Percentage of Participants With A1C at Goal (<6.5%) at Week 20
Description: Glycated hemoglobin (A1C) is a blood marker used to report average blood glucose levels over prolonged periods of time. Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100. Percentage of participants with A1C at goal (<6.5%) at Week 20 was presented.
Time Frame: Week 20
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled | Metformin and Metformin XR Pooled
Number analyzed (Participants) | 107 | 113
Percentage of participants | 29.0 | 20.4
Statistical Analysis 1: Comparison: Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled vs Metformin and Metformin XR Pooled; The percentage of participants with A1C at the A1C goal (<6.5%) in the arm "Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled" is compared against that of "Metformin and Metformin XR Pooled." For estimating the treatment difference, when the A1C result for a participant at Week 20 was not available, a multiple imputation method was used to impute whether the participant had met the goal; Test type: Superiority; p = 0.049, Miettinen and Nurminen; Difference in Percentage = 12.2, 95% CI 2-sided [0.0 to 24.8]

11. Secondary Outcome: Percentage of Participants With A1C at Goal (<7.0%) at Week 54
Description: Glycated hemoglobin (A1C) is a blood marker used to report average blood glucose levels over prolonged periods of time. Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100. Percentage of participants with A1C at goal (<7.0%) at Week 54 was presented.
Time Frame: Week 54
Population: The analysis population includes all randomized participants who received ≥1 dose of study medication and continued in the study beyond Week 20. As defined in the protocols, these analyses were conducted in participants pooled from protocols MK-0431A-170 and MK-0431A-289, pooled according to receipt of experimental drug or placebo comparator.
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled | Metformin and Metformin XR Pooled
Number analyzed (Participants) | 70 | 77
Percentage of participants | 31.4 | 27.3

12. Secondary Outcome: Percentage of Participants With A1C at Goal (<6.5%) at Week 54
Description: Glycated hemoglobin (A1C) is a blood marker used to report average blood glucose levels over prolonged periods of time. Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100. Percentage of participants with A1C at goal (<6.5%) at Week 54 was presented.
Time Frame: Week 54
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled | Metformin and Metformin XR Pooled
Number analyzed (Participants) | 70 | 77
Percentage of participants | 18.6 | 19.5

13. Secondary Outcome: Percentage of Participants Initiating Glycemic Rescue Therapy by Week 20
Description: Percentage of participants who initiated glycemic rescue therapy prior to Week 20 was reported.
Time Frame: Up to Week 20
Population: The analysis population includes all randomized participants who received ≥1 dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin/Metformin | Metformin | Sitagliptin/Metformin XR | Metformin XR | Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled | Metformin and Metformin XR Pooled
Number analyzed (Participants) | 62 | 62 | 45 | 51 | 107 | 113
Percentage of participants | 3.2 | 19.4 | 4.4 | 13.7 | 3.7 | 16.8
Statistical Analysis 1: Comparison: Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled vs Metformin and Metformin XR Pooled; The percentage of participants initiating glycemic rescue therapy in the arm "Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled" is compared against that of "Metformin and Metformin XR Pooled."; Test type: Superiority; p = 0.002, Log-Rank Test; Kaplan-Meier Difference in Percentage = -13.2, 95% CI 2-sided [-21.1 to -5.3]

14. Secondary Outcome: Percentage of Participants Initiating Insulin Glargine During Weeks 20-54
Description: Percentage of participants who initiated insulin glargine therapy from Weeks 20 through 54 was reported.
Time Frame: Week 20 up to Week 54
Population: The analysis population includes all randomized participants who received ≥1 dose of study medication and continued in the study beyond Week 20 without initiating glycemic rescue therapy before Week 20. As defined in the protocols, these analyses were on participants pooled from protocols MK-0431A-170 and -289, pooled by receipt of drug or placebo.
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled | Metformin and Metformin XR Pooled
Number analyzed (Participants) | 66 | 64
Percentage of participants | 22.7 | 26.6

15. Other Pre Specified Outcome: Baseline A1C
Description: Glycated hemoglobin (A1C) is a blood marker used to report average blood glucose levels over prolonged periods of time. Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100.
Time Frame: Baseline
Population: The analysis population includes all randomized participants who received ≥1 dose of study medication and had a baseline measurement of A1C. Baseline A1C data for non-pooled arms are listed in the Baseline Characteristics module.
Measure: Mean (Standard Deviation); unit: Percentage of glycated hemoglobin
Arm/Group | Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled | Metformin and Metformin XR Pooled
Number analyzed (Participants) | 107 | 113
Percentage of glycated hemoglobin | 7.96 (1.11) | 8.06 (1.07)

ADVERSE EVENTS:
Time Frame: Up to 56 weeks for non-serious adverse events. Up to approximately 76 weeks for serious adverse events. Up to approximately 78 weeks for all-cause mortality.
Description: "Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled" = "Sitagliptin/Metformin" plus "Sitagliptin/Metformin XR." "Metformin and Metformin XR Pooled" = "Metformin" plus "Metformin XR."
  Non-serious and serious adverse events are recorded for all treated participants.
  All-cause mortality is recorded for all randomized participants.
Arm/Group | Sitagliptin/Metformin | Metformin | Sitagliptin/Metformin XR | Metformin XR | Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled | Metformin and Metformin XR Pooled
All-Cause Mortality (participants affected / at risk) | 1/62 | 0/62 | 0/47 | 0/51 | 1/109 | 0/113
Serious Adverse Events (participants affected / at risk) | 4/62 | 3/62 | 3/45 | 3/51 | 7/107 | 6/113
Other Adverse Events (participants affected / at risk) | 34/62 | 40/62 | 30/45 | 36/51 | 64/107 | 76/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin/Metformin (N=62) | Metformin (N=62) | Sitagliptin/Metformin XR (N=45) | Metformin XR (N=51) | Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled (N=107) | Metformin and Metformin XR Pooled (N=113)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Type I hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
H1N1 influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin/Metformin (N=62) | Metformin (N=62) | Sitagliptin/Metformin XR (N=45) | Metformin XR (N=51) | Sitagliptin/Metformin and Sitagliptin/Metformin XR Pooled (N=107) | Metformin and Metformin XR Pooled (N=113)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (4) | 4 (4) | 4 (4) | 6 (6) | 8 (8)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 2 (2) | 0 (0) | 3 (4) | 1 (2) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 4 (4) | 1 (1) | 3 (10) | 8 (9) | 7 (14)
Nausea (Gastrointestinal disorders) | 2 (5) | 5 (5) | 4 (6) | 2 (3) | 6 (11) | 7 (8)
Gastroenteritis (Infections and infestations) | 5 (6) | 3 (3) | 3 (3) | 2 (2) | 8 (9) | 5 (5)
Influenza (Infections and infestations) | 1 (1) | 4 (5) | 2 (3) | 3 (5) | 3 (4) | 7 (10)
Nasopharyngitis (Infections and infestations) | 7 (11) | 7 (7) | 1 (2) | 2 (3) | 8 (13) | 9 (10)
Pharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 5 (6) | 2 (2) | 8 (9)
Upper respiratory tract infection (Infections and infestations) | 9 (11) | 6 (8) | 5 (9) | 3 (5) | 14 (20) | 9 (13)
Urinary tract infection (Infections and infestations) | 0 (0) | 5 (6) | 3 (3) | 1 (1) | 3 (3) | 6 (7)
Alanine aminotransferase increased (Investigations) | 2 (3) | 3 (3) | 3 (3) | 3 (3) | 5 (6) | 6 (6)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 1 (1) | 3 (3) | 1 (1) | 6 (6) | 2 (2)
Blood glucose increased (Investigations) | 3 (4) | 0 (0) | 2 (2) | 3 (5) | 5 (6) | 3 (5)
Creatinine renal clearance increased (Investigations) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Urine albumin/creatinine ratio increased (Investigations) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 4 (5) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 5 (6) | 3 (3) | 4 (4) | 6 (6) | 9 (10)
Hypoglycaemia (Metabolism and nutrition disorders) | 10 (106) | 6 (15) | 9 (70) | 10 (45) | 19 (176) | 16 (60)
Headache (Nervous system disorders) | 3 (4) | 8 (10) | 2 (4) | 10 (15) | 5 (8) | 18 (25)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4) | 3 (3) | 2 (2) | 5 (5) | 5 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (6) | 5 (5) | 2 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/47/NCT01760447/Prot_SAP_000.pdf